CLINICAL TRIAL: NCT01469611
Title: A Phase 1b Dose Escalation Study of JX-594 (Thymidine Kinase-Inactivated Vaccinia Virus Plus GM-CSF) Administered by Biweekly (Every Two Weeks) Intravenous Infusion in Patients With Metastatic, Refractory Colorectal Carcinoma
Brief Title: A Trial of JX-594 in Refractory Colorectal Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Young Suk Park, Professor of Medicine, Sungkyunkwan University School of Medicine, Department of Hematology and Oncology, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC IRB 2009-06-055
Record Dates: First submitted 2011-11-07; First posted 2011-11-10 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Colorectal Carcinoma
Keywords: advanced/metastatic colorectal carcinoma
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- JX-594 (Experimental): Infusion Procedure:JX-594 will be administered on the designated treatment days at a dose of either 1 x 106, 1 x 107 or 3 x 107 pfu per kg. Virus infusion should occur over 60 minutes (+/- 5 minutes). The final infusion volume of virus plus diluent will be approximately 250 mL.
  Interventions: Biological: JX-594

INTERVENTIONS:
Biological: JX-594 — Infusion Procedure:JX-594 will be administered on the designated treatment days at a dose of either 1 x 106, 1 x 107 or 3 x 107 pfu per kg. Virus infusion should occur over 60 minutes (+/- 5 minutes). The final infusion volume of virus plus diluent will be approximately 250 mL.

SUMMARY:
The purpose of this study is to:

* determine the maximally-tolerated dose (MTD) and/or maximum-feasible dose (MFD) of JX-594 administered by biweekly intravenous (IV) infusion.
* determine the safety of JX-594(TK- GM-CSF+ Wyeth strain vaccinia) administered by biweekly IV infusion.

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, dose-escalation trial in patients with advanced colorectal carcinoma (CRC) that have failed both oxaliplatin based and irinotecan based prior chemotherapy regimens for metastatic disease. Patients will receive treatment at one of three dose levels in a sequential dose-escalating design.

Three patients will be treated at each dose level unless a dose-limiting toxicity (DLT) is observed. Enrollment will proceed to the next dose level if 0 of 3 patients experiences a DLT; if one of the first 3 patients experiences a DLT, additional patients will be enrolled until a second patient experiences a DLT (which defines the toxic dose) or until six total patients have been treated at that dose level, whichever comes first. If a second DLT is not experienced within that cohort, dose escalation may continue.

Patients will be enrolled a minimum of 14 days after the first treatment of the immediately preceding patient for the first patient in any cohort or all remaining patients in a cohort with DLT.

If 2 DLTs are observed within a cohort, enrollment into the cohort will cease and the dose level immediately preceding that dose will be determined to be the MTD. Regulatory Authorities and the IRB will be notified as required if any patient dies within 28 days of product administration due to a serious and unexpected ADR that is determined by the Investigator to be possibly or probably related to JX-594.

Once the MTD and/or MFD is defined, an additional 3-6 patients may be enrolled at that dose level. Note: once the MTD and/or MFD is defined, treatment of additional patients at this dose level will no longer require inter-patient delays of 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed, advanced/metastatic colorectal carcinoma
* Failed both oxaliplatin and irinotecan based regimens for advanced/metastatic disease (tumor progression on or within 3 months of treatment completion)
* Erbitux therapy resistant: Ras mutant tumor status, and/or failed Erbitux therapy (tumor progression on or within 3 months of treatment completion or Erbitux treatment not indicated due to lack of epidermal growth factor (EGFR) expression)
* At least one measurable tumor mass by PET-CT/CT/MRI (lesion that can accurately be measured in at least one dimension with longest diameter > 1 cm)
* Expected survival for approximately 12 weeks or longer
* Karnofsky Performance Score (KPS) ≥ 70
* Age ≥18 years
* WBC ≥ 3,500 cells/mm3 and ≤ 50,000 cells/mm3
* ANC ≥ 1,500 cells/mm3
* Hemoglobin ≥ 10 g/dL (transfusion allowed)
* Platelet count ≥ 100,000 plts/mm3
* Total bilirubin ≤ 1.5 ULN
* AST, ALT ≤2.5 ULN (if liver metastases(+): AST,ALT ≤5.0 x ULN)
* Serum chemistries within normal limits (WNL) or Grade 1 (excluding alkaline phosphatase) - If patients are diabetic or have a screening random glucose > 160 mg/dL, a fasting glucose must be done and patients must be WNL or Grade 1 in order to be eligible for the study.

Exclusion Criteria:

* Significant immunodeficiency due to underlying illness (e.g. HIV/AIDS) and/or medication (e.g. systemic corticosteroids)
* Known myeloproliferative disorders requiring systemic therapy
* History of exfoliative skin condition (e.g. eczema or ectopic dermatitis) requiring systemic therapy
* History of acquiring opportunistic infections.
* Tumor(s) invading a major vascular structure (e.g. carotid artery)
* Tumor(s) in location that would potentially result in significant clinical adverse effects if post-treatment tumor swelling were to occur (e.g. tumors impinging on the upper airway or affecting biliary tract drainage, etc.)
* Clinically significant and/or rapidly accumulating ascites, peri-cardial and/or pleural effusions
* Severe or unstable cardiac disease, including (for example) coronary artery disease requiring increased doses of anti-anginal mediation and/or coronary angioplasty (including stent placement) within the preceding 24 months
* Current, known CNS malignancy (history of completely resected or irradiated brain metastases by WBRT or stereotactic radiosurgery allowed)
* Received anti-cancer therapy within 4 weeks prior to first treatment (6 weeks in case of mitomycin C or nitrosoureas)
* Use of anti-viral, anti-platelet, or anti-coagulation medication [Patients who discontinue such medications within 7 days prior to first treatment may be eligible for this study.] Low dose aspirin (approximately 81 mg) allowed.
* Pulse oximetry O2 saturation <90% at rest
* Experienced a severe systemic reaction or side-effect as a result of a previous smallpox vaccination

Household contact exclusions:

* Women who are pregnant or nursing an infant
* Children < 12 months old
* People with skin disease (e.g. eczema, atopic dermatitis, and related diseases Immunocompromised hosts (severe deficiencies in cell-mediated immunity, including AIDS, organ transplant recipients, hematologic malignancies)Patients with household contacts meeting any of the above criteria will be excluded unless alternate living arrangements can be made during the patient's dosing period and for at least 7 days following the last dose of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Determine the maximally-tolerated dose | 18 months
Determine the maximum-feasible dose | 18months

CONTACTS AND LOCATIONS:
Overall Officials: Young suk park, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea